CLINICAL TRIAL: NCT06834308
Title: The Effect of Transcutaneous Electrical Nerve Stimulation on Exercise-Induced Pain in Women Living With Fibromyalgia
Brief Title: TENS Therapy to Reduce Exercise-Induced Pain in Women With Fibromyalgia
Acronym: TENSXFibro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor at Faculty of Medecine and Health Sciences of Université de Sherbrooke, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-5394
Record Dates: First submitted 2025-02-12; First posted 2025-02-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; TENS; Exercise; Exercise-Induced Pain; Sham; Conventional; Women
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding assessment: Participants' treatment expectations (before and after the first TENS application) will be used as an indicator of blinding success. The outcome assessor's blinding will be assessed by asking them to guess the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional TENS with Resistance Exercise (Experimental): Conventional TENS will be administered using a 2-channel TENS unit (Biomed 2000XL) and carbon electrodes. Electrodes will be placed on the area identified by the participant as most painful (loco dolenti). The TENS parameters will be set to conventional stimulation (100 Hz, 60 ms), with the intensity adjusted to produce a strong paresthesia sensation without causing pain. TENS will be applied for 10 minutes before the first set and maintained throughout the exercise sets.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Sham TENS with Resistance Exercise (Sham Comparator): The sham TENS procedure will mimic the conventional TENS procedure, but the modified TENS device will not deliver electrical stimulation. Participants will be blinded to the intervention they will receive and will be told they could receive 2 types of TENS.
  Interventions: Device: SHAM Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Conventional TENS (100 Hz, 60 ms pulse width) will be applied for 10 minutes prior to and during resistance exercise (2 sets of 10 reps at 60% 1RM leg press). TENS' intensity will be adjusted to produce strong paresthesia without pain. Electrodes will be placed on participant-identified most painful area. Resistance exercise will consist of two sets of ten repetition with 1 min rest
  Arms: Conventional TENS with Resistance Exercise
Device: SHAM Transcutaneous electrical nerve stimulation (TENS) — The participants will be able to see the same parameters as the conventional TENS (100 Hz, 60 ms pulse width) on the screen, but there will be no actual stimulation. Sham TENS will be applied for 10 minutes prior to and during resistance exercise (2 sets of 10 reps at 60% 1RM leg press). TENS' intensity will be adjusted to 4Hz for all participants in the Sham arm. Electrodes will be placed on participant-identified most painful area. Resistance exercise will consist of two sets of ten repetition with 1 min rest
  Arms: Sham TENS with Resistance Exercise

SUMMARY:
The goal of this clinical trial is to evaluate the short-term (24-hour) effect of conventional transcutaneous electrical nerve stimulation (TENS) compared to Sham TENS on pain induced by resistance training in women with fibromyalgia. The main questions it aims to answer are:

1. Can conventional TENS effectively reduce pain intensity and unpleasantness during and after a resistance training session in women with fibromyalgia?
2. Is there a significant difference between the effects of conventional TENS and Sham TENS on exercise-induced pain in this population? Researchers will compare a conventional TENS group to a Sham TENS group to see if active TENS application during and after resistance training sessions leads to reduced pain levels and improved pain perception.

Participants will:

* Undergo a supervised resistance training session
* Receive either conventional TENS or ShamTENS treatment during and after exercise
* Complete pain assessments, measuring both intensity and unpleasantness, before, during, and up to 24 hours after exercise sessions

DETAILED DESCRIPTION:
Study Design

Randomization with minimization will be performed using MinimPy software to ensure group balance, considering the following factors:

* Pain intensity, assessed using a pain scale (0-10)
* Fibromyalgia severity, assessed using the Fibromyalgia Impact Questionnaire
* Age

Participants will be informed that different types of TENS stimulation may or may not produce a sensation, and this does not impact treatment effectiveness.

Resistance Exercise Protocol The resistance training protocol involves a leg press exercise performed at a 90° starting angle. Participants will undergo a familiarization period, a warm-up, and a repetitions-to-failure (RTF) test to determine their 5-repetition maximum (RM). The Epley equation will be used to predict the 1RM. Participants will then perform two sets of 10 repetitions at 60% of their estimated 1RM, with a 1-minute rest between sets. A kinesiologist will supervise the training session.

Data Collection

Baseline Assessments:

Demographic information (age, gender identity, height, weight, medication) Physical activity level (Physical Activity Questionnaire for Adults) Fibromyalgia severity (Fibromyalgia Impact Questionnaire) Kinesiophobia (Tampa Scale of Kinesiophobia) Treatment expectations (Numerical scale from -100 to 100) Blood pressure Repetitions to Failure Test (RTF)

Participants will also complete a digital logbook via REDCap to record their pain levels at the end of the day and 24 hours post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* Be 40 years of age or older.
* Have a diagnosis of fibromyalgia.
* Experience persistent pain in the lumbo-pelvic and lower limb region with an intensity ≥ 3/10 on a numerical scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable).
* Refrain from consuming caffeine and analgesics 6 hours before the experiment, and refrain from smoking cigarettes 2 hours before the experiment.

Exclusion Criteria:

* Are physically active prior to the start of the study, i.e., they meet the recommendations of 150 minutes per week of moderate to vigorous intensity activity or practice 2 times 30 minutes of muscle-strengthening exercises per week for 2 months.
* Suffer from poorly controlled cardiovascular diseases.
* Have one or more contraindications to physical activity
* Have one or more contraindications to TENS
* Have already participated in a research project involving TENS or used a TENS device in the past 10 years.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | At baseline, immediately post-exercise, 15 minutes post-exercise, end of the day of the visit, and 24 hours post-exercise.
  Pain intensity will be measured using a Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents "no pain" and 10 represents "worst pain imaginable."

SECONDARY OUTCOMES:
Unpleasantness of pain | At baseline, immediately post-exercise, 15 minutes post-exercise, end of the day of the visit, and 24 hours post-exercise.
  The unpleasantness of pain will be measured using a Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents "pain is not unpleasant" and 10 represents "pain is the most unpleasant imaginable."

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided